CLINICAL TRIAL: NCT03065751
Title: Prospective, Randomized, Multicenter, Open-label, Controlled, Parallel-group Trial Investigating the Efficacy of add-on Plasma-exchange as an Adjunctive Strategy Against Septic Shock
Brief Title: Plasmaexchange in Early Septic Shock
Acronym: EXCHANGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2786-2015
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPE (Active Comparator)
  Interventions: Device: Plasmaexchange
- Kontroll (No Intervention)

INTERVENTIONS:
Device: Plasmaexchange — TPE against fresh frozen plasma
  Arms: TPE

SUMMARY:
Sepsis is defined by the occurrence of a systemic inflammatory response syndrome (SIRS) in the context of infection. Unfortunately, its incidence appears to be rising, and the mortality of septic shock remains extraordinary high (> 60%). Death in sepsis arises from shock and multi organ dysfunction that are - at least in part - triggered by an inadequate response of the host's immune system to the infection. Given the injurious role of 1) this overwhelming immune response and 2) the consumption of protective plasmatic factors (e.g. vWF cleaving proteases, hemostatic factors etc.) while the disease is progressing the investigators hypothesize that early therapeutic plasma exchange (TPE) in the most severely ill individuals might improve hemodynamics, oxygenation and ultimately survival. This therapeutic strategy combines 2 major aspects in 1 procedure: 1. removal of harmful circulating molecules and 2. replacement of protective plasma proteins. The investigators designed the EXCHANGE trial to analyze in a randomized fashion the benefit of TPE as an add-on treatment to state of the art standard sepsis care. Only patients with early septic shock (< 12 hrs) and high catecholamine doses (noradrenaline > 0.4 ug/kg bodyweight/min) will be included. Those in the treatment group will receive 3 TPEs within three consecutive days. The primary outcome is 28-day all cause mortality. To show an assumed reduction from 60% to 45% in the experimental group, a sample size of 173 patients per group has been calculated. The overall sample size is therefore n=346. The recruitment period is 3 years (+3 months observation) and will be performed in 11 national centers in Germany. Secondary endpoints (including hemodynamics, oxygenation, coagulation, and microcirculation) will be assessed on day 1, 2, 3 before and after TPE and on day 4, 5, 7 and 14.

Project management and data monitoring will be organized by the Hanover Clinical Trial Center and biostatistics including a web-based randomization will be performed by the Institute of biometrics (Prof. Koch) at Hannover Medical School.

The investigators hope to demonstrate a potential benefit of an additive treatment approach to improve the outcome of patients suffering from an under-recognized but deadly disease.

ELIGIBILITY:
Inclusion Criteria:

* Onset of septic shock within less than 12 hrs
* Noradrenaline dose of ≥ 0.4 ug/kg/min bodyweight (target MAD ≥ 65 mmHg) ≥ 30 min

Exclusion Criteria:

* Age<18 years and > 80 years
* Pregnancy
* Known history of transfusion reactions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days
  Overall mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
pre-defined substudies with primary responsibilities for each individual center

REFERENCES:
- [Derived] Stahl K, Schmidt JJ, Seeliger B, Schmidt BMW, Welte T, Haller H, Hoeper MM, Budde U, Bode C, David S. Effect of therapeutic plasma exchange on endothelial activation and coagulation-related parameters in septic shock. Crit Care. 2020 Mar 2;24(1):71. doi: 10.1186/s13054-020-2799-5. PMID 32122366
- [Derived] Knaup H, Stahl K, Schmidt BMW, Idowu TO, Busch M, Wiesner O, Welte T, Haller H, Kielstein JT, Hoeper MM, David S. Early therapeutic plasma exchange in septic shock: a prospective open-label nonrandomized pilot study focusing on safety, hemodynamics, vascular barrier function, and biologic markers. Crit Care. 2018 Oct 30;22(1):285. doi: 10.1186/s13054-018-2220-9. PMID 30373638